CLINICAL TRIAL: NCT01558401
Title: Effects of an Adapted Physical Activity Program on the Physical Condition of Elderly Women: an Analysis of Efficiency
Brief Title: Efficiency of Physical Activity on the Physical Condition of Elderly Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sao Carlos (Other)
Responsible Party: Principal Investigator, Francisco Alburquerque, Ph.D., Assistant Professor, Universidade Federal de Sao Carlos
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Ethics Committe UFSCar Nº104/4
Record Dates: First submitted 2012-03-14; First posted 2012-03-20 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Aging
Keywords: physical activity; elderly; women; efficiency
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Physical activity program Group (Experimental): The physical activity program consists of 123 sessions over 52 weeks. The initial assessment is followed by 12 weeks of physical activity. After this ten-week period, a second assessment is performed, followed by 3 weeks of rest. This is followed by a further 17 weeks of activities, 4 weeks of activities followed by 4 weeks of rest. Finally, there were 12 more weeks of activities.
  Interventions: Other: Physical activity program

INTERVENTIONS:
Other: Physical activity program — The activities are done in groups of no more than 25 individuals; these activities are standardized and agreed upon by the research team, which hold monthly meetings to conduct the study. Each physical activity session consists of 8-10 minutes of exercises aimed at stretching the major muscle groups (pectoral muscles, latissimus dorsi, cervical paravertebral, and posterior and anterior thigh muscles); 9 minutes of aerobic endurance activity (march/fast walk); 7-10 minutes of adapted strength exercises, power, and endurance training; 14-16 minutes of coordination, agility, and flexibility exercises, and 5-7 minutes of respiratory and relaxation exercises.

SUMMARY:
The purpose of this study was to identify the effects and the efficiency of an adapted physical activity program as regards the physical condition of older Brazilian women.

DETAILED DESCRIPTION:
Although physical activity programs for the elderly have proved to be able to curb harmful changes due to ageing, not all programs show the same effectiveness, even though they are generally regarded as being effective. The existence of a wide variety of programs calls for debate about their outcomes.

Specific research tools and designs can assist in identifying not only program effectiveness but also program efficiency and use in terms of a better physical performance of subjects on carrying out exercises with less effort, influenced by multiple factors, one of them being adherence to the program. These analyses allow the influence of efficiency and the factors that determine it or are associated with it to be tested, and can provide classifications and subgroups to which interventions should be adapted if they are to offer the best service to them in the short and medium term.

ELIGIBILITY:
Inclusion Criteria:

* 60 or more years
* participants of an Adult Revitalization Program in São Carlos (São Paulo State - Brazil)

Exclusion Criteria:

* physical characteristics and previous health problems that might hinder their participation in the program activities.
* adherence to the program sessions lower than 75%.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-04; Primary Completion 2011-04 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Efficiency Data Envelopment Analysis (DEA) | 1 year
  Data Envelopment Analysis (DEA) is a test of operational investigation It was used to determine the relative efficiency of the older women, considered Decision Making Units (DMU). This analysis supports the hypothesis that the outputs do not need to be proportional to the inputs.

SECONDARY OUTCOMES:
Grip strength | 1 year
  Grip strength was measured using a Sammons Preston Swedley-Type hand dynamometer (Jamar® Bolingbrook IL, 60440). The test was performed three times on the dominant upper limb at 10-second intervals between each run. The grip strength assigned to each participant was the highest of the three values measured. Subjects were guided to hold the grip meter during exhalation without performing the Valsalva maneuver; they were encouraged verbally throughout the test.
Sit-and-Reach Test | 1 year
  The Sit-and-Reach Test was employed to evaluate the participants' flexibility of the posterior trunk and lower limbs. The movement was performed three times. The flexibility assigned to subjects was the highest value measured.
Static balance | 1 year
  Static balance was verified by the One-Leg Stance Test with eyes open31. The subjects gazed at a fixed point two meters away for no more than 30 seconds, with one leg bent at the knee. The test was done three times with open and closed eyes and for both legs, taking into account for each condition (open or closed eyes) the mean value of the measures.
Dynamic balance | 1 year
  Dynamic balance was evaluated by the Maximum Gait Velocity (MGV). The subjects were instructed to walk along a 33.3cm-wide and 3.33m-long band painted on the floor in the shortest possible time. The test was performed three times. The dynamic balance value assigned to each subject was the mean time walking along the band.
VO2max | 1 year
  The Rockport 1-Mile Walk Test was used to determine the subjects' physical condition estimated by the VO2max

CONTACTS AND LOCATIONS:
Overall Officials: José R. Rebelatto, Ph.D., Principal Investigator — Universidade Federal de Sao Carlos
Locations (1):
- Universidade Federal de Sao Carlos, São Carlos, São Paulo, Brazil

REFERENCES:
- [Background] Gillespie LD, Robertson MC, Gillespie WJ, Lamb SE, Gates S, Cumming RG, Rowe BH. Interventions for preventing falls in older people living in the community. Cochrane Database Syst Rev. 2009 Apr 15;(2):CD007146. doi: 10.1002/14651858.CD007146.pub2. PMID 19370674
- [Background] Conn VS, Minor MA, Burks KJ, Rantz MJ, Pomeroy SH. Integrative review of physical activity intervention research with aging adults. J Am Geriatr Soc. 2003 Aug;51(8):1159-68. doi: 10.1046/j.1532-5415.2003.51365.x. PMID 12890083
- [Background] Laine J, Finne-Soveri UH, Bjorkgren M, Linna M, Noro A, Hakkinen U. The association between quality of care and technical efficiency in long-term care. Int J Qual Health Care. 2005 Jun;17(3):259-67. doi: 10.1093/intqhc/mzi032. Epub 2005 Mar 23. PMID 15788463
- [Background] Greve P, Wanderley FDS, Rebelatto JR. The effects of periodic interruptions of physical activities on the physical capacities of adult active women. Arch Gerontol Geriatr. 2009 Sep-Oct;49(2):268-271. doi: 10.1016/j.archger.2008.09.009. Epub 2008 Nov 6. PMID 18992949
- [Background] Vogel T, Brechat PH, Lepretre PM, Kaltenbach G, Berthel M, Lonsdorfer J. Health benefits of physical activity in older patients: a review. Int J Clin Pract. 2009 Feb;63(2):303-20. doi: 10.1111/j.1742-1241.2008.01957.x. PMID 19196369
- [Derived] Alburquerque-Sendin F, Barberio-Mariano E, Brandao-Santana N, Rebelatto DA, Rebelatto JR. Effects of an adapted physical activity program on the physical condition of elderly women: an analysis of efficiency. Rev Bras Fisioter. 2012 Jul-Aug;16(4):328-36. doi: 10.1590/s1413-35552012005000025. Epub 2012 Jun 14. PMID 22699693